CLINICAL TRIAL: NCT02646488
Title: Using Practice Facilitation in Primary Care Settings to Reduce Risk Factors for Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 14-02042
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Disease; High Blood Pressure
Keywords: cholesterol; smoking; aspirin; chronic care model
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Smoking | interventions — Chronic Care Model

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cluster 1 (Active Comparator): Consists of 80 sites chosen by block randomization in four waves every three months (80 in the first three waves and 60 in the last wave).
  Interventions: Behavioral: Million Hearts ABCS 6 Months; Behavioral: Standard Care Regimen 9 Months; Behavioral: Standard Care Regimen 12 Months; Behavioral: Standard Care Regimen 15 Months; Behavioral: Standard Care Regimen 18 Months; Behavioral: Follow Up Post Intervention 21 Months; Behavioral: Follow Up Post Intervention 24 Months
- Cluster 2 (Active Comparator): Consists of 80 sites chosen by block randomization in four waves every three months (80 in the first three waves and 60 in the last wave).
  Interventions: Behavioral: Million Hearts ABCS 6 Months; Behavioral: Million Hearts ABCS 9 Months; Behavioral: Standard Care Regimen 12 Months; Behavioral: Standard Care Regimen 15 Months; Behavioral: Standard Care Regimen 18 Months; Behavioral: Standard Care Regimen 21 Months; Behavioral: Follow Up Post Intervention 24 Months; Behavioral: Follow Up Post Intervention 27 Months
- Cluster 3 (Active Comparator): Consists of 80 sites chosen by block randomization in four waves every three months (80 in the first three waves and 60 in the last wave).
  Interventions: Behavioral: Million Hearts ABCS 6 Months; Behavioral: Million Hearts ABCS 9 Months; Behavioral: Million Hearts ABCS 12 Months; Behavioral: Standard Care Regimen 15 Months; Behavioral: Standard Care Regimen 18 Months; Behavioral: Standard Care Regimen 21 Months; Behavioral: Standard Care Regimen 24 Months; Behavioral: Follow Up Post Intervention 27 Months; Behavioral: Follow Up Post Intervention 30 Months
- Cluster 4 (Active Comparator): Consists of 80 sites chosen by block randomization in four waves every three months (80 in the first three waves and 60 in the last wave).
  Interventions: Behavioral: Million Hearts ABCS 6 Months; Behavioral: Million Hearts ABCS 9 Months; Behavioral: Million Hearts ABCS 12 Months; Behavioral: Million Hearts ABCS 15 Months; Behavioral: Standard Care Regimen 18 Months; Behavioral: Standard Care Regimen 21 Months; Behavioral: Standard Care Regimen 24 Months; Behavioral: Standard Care Regimen 27 Months; Behavioral: Follow Up Post Intervention 30 Months; Behavioral: Follow Up Post Intervention 33 Months

INTERVENTIONS:
Behavioral: Million Hearts ABCS 6 Months — The ABCS refer to the following: Aspirin in high-risk individuals (A), Blood pressure control and management (B), Cholesterol management (C), and Smoking cessation (S).
  Other Names: Chronic Care Model
Behavioral: Million Hearts ABCS 9 Months — The ABCS refer to the following: Aspirin in high-risk individuals (A), Blood pressure control and management (B), Cholesterol management (C), and Smoking cessation (S).
  Arms: Cluster 2; Cluster 3; Cluster 4
Behavioral: Million Hearts ABCS 12 Months — The ABCS refer to the following: Aspirin in high-risk individuals (A), Blood pressure control and management (B), Cholesterol management (C), and Smoking cessation (S).
  Arms: Cluster 3; Cluster 4
Behavioral: Million Hearts ABCS 15 Months — The ABCS refer to the following: Aspirin in high-risk individuals (A), Blood pressure control and management (B), Cholesterol management (C), and Smoking cessation (S).
  Arms: Cluster 4
Behavioral: Standard Care Regimen 9 Months
  Arms: Cluster 1
Behavioral: Standard Care Regimen 12 Months
  Arms: Cluster 1; Cluster 2
Behavioral: Standard Care Regimen 15 Months
  Arms: Cluster 1; Cluster 2; Cluster 3
Behavioral: Standard Care Regimen 18 Months
Behavioral: Standard Care Regimen 21 Months
  Arms: Cluster 2; Cluster 3; Cluster 4
Behavioral: Standard Care Regimen 24 Months
  Arms: Cluster 3; Cluster 4
Behavioral: Standard Care Regimen 27 Months
  Arms: Cluster 4
Behavioral: Follow Up Post Intervention 21 Months
  Arms: Cluster 1
Behavioral: Follow Up Post Intervention 24 Months
  Arms: Cluster 1; Cluster 2
Behavioral: Follow Up Post Intervention 27 Months
  Arms: Cluster 2; Cluster 3
Behavioral: Follow Up Post Intervention 30 Months
  Arms: Cluster 3; Cluster 4
Behavioral: Follow Up Post Intervention 33 Months
  Arms: Cluster 4

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness of practice facilitation as a quality improvement strategy for implementing the Million Hearts' ABCS treatment guidelines for reducing cardiovascular disease (CVD) among high-risk patients who receive care in primary care practices in New York City. The ABCS refer to the following: Aspirin in high-risk individuals (A), Blood pressure control and management (B), Cholesterol management (C), and Smoking cessation (S). The long-term goal is to create a robust infrastructure to disseminate and implement evidence based practice guidelines (EBPG) findings in primary care practices and improve practices' capacity to receive and implement other EBPG findings in the future.

ELIGIBILITY:
Inclusion Criteria:

Provider and staff eligibility inclusion criteria.

* Eligibility includes working full or part time at the study site.

Stakeholder eligibility inclusion criteria.

* Steering committee members or other key stakeholder from the following groups: Health Plan Chief Medical Officer, State health officials in the Chronic Disease Program, and leadership from relevant national associations (American Heart Association), members of Advisory Board of CHCANYS (these are physician leaders).

Patient eligibility inclusion criteria:

* at least one of the ABCS risk factors for CVD (i.e., hypertension, hyperlipidemia, eligible for aspirin and/or is a current smoker)
* must have received care at the clinic for at least 12 months
* Patients eligible for aspirin are those with a documented ICD-9 code for ischemic vascular disease in the last 12 months. Similarly, patients with a diagnosis of hypertension and/or hyperlipidemia will have a documented ICD-9 code for the targeted risk factor
* Smokers will be identified by a documented ICD-9 code, prescription for a cessation medication in the last 12 months or documentation in the chart (e.g. meaningful use measure) during the last 12 months (see outcome measures)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with documented use of aspirin or other antithrombotic. | 18 Months
Percentage of patients who had a diagnosis of hypertension (HTN) and whose blood pressure (BP) was adequately controlled | 18 Months
Percentage of patients who had a fasting lipoprotein (LDL) test performed and whose risk-stratified fasting LDL is at or below the recommended low density lipoprotein (LDL) goal | 18 Months
Change in the percentage of patients who had a low density lipoprotein (LDL) test who are prescribed a recommended dose of statin based on risk status if indicated. | 18 Months
Percentage of patients who were screened about tobacco use one or more times within 24 months AND who received cessation counseling intervention if identified as a tobacco user. | 24 Months

SECONDARY OUTCOMES:
Percentage of patients aged 18 through 85 years of age who had a diagnosis of hypertension (HTN) who are prescribed recommended medications, if indicated. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Gold HT, Siman N, Cuthel AM, Nguyen AM, Pham-Singer H, Berry CA, Shelley DR. A practice facilitation-guided intervention in primary care settings to reduce cardiovascular disease risk: a cost analysis. Implement Sci Commun. 2021 Feb 6;2(1):15. doi: 10.1186/s43058-021-00116-x. PMID 33549152
- [Derived] Berry CA, Nguyen AM, Cuthel AM, Cleland CM, Siman N, Pham-Singer H, Shelley DR. Measuring Implementation Strategy Fidelity in HealthyHearts NYC: A Complex Intervention Using Practice Facilitation in Primary Care. Am J Med Qual. 2021 Jul-Aug 01;36(4):270-276. doi: 10.1177/1062860620959450. PMID 32964719
- [Derived] Shelley DR, Gepts T, Siman N, Nguyen AM, Cleland C, Cuthel AM, Rogers ES, Ogedegbe O, Pham-Singer H, Wu W, Berry CA. Cardiovascular Disease Guideline Adherence: An RCT Using Practice Facilitation. Am J Prev Med. 2020 May;58(5):683-690. doi: 10.1016/j.amepre.2019.12.013. Epub 2020 Feb 14. PMID 32067871
- [Derived] Gepts T, Nguyen AM, Cleland C, Wu W, Pham-Singer H, Shelley D. Accounting for Blood Pressure Seasonality Alters Evaluation of Practice-Level Blood Pressure Control Intervention. Am J Hypertens. 2020 Mar 13;33(3):220-222. doi: 10.1093/ajh/hpz179. PMID 31711219
- [Derived] Shelley DR, Ogedegbe G, Anane S, Wu WY, Goldfeld K, Gold HT, Kaplan S, Berry C. Testing the use of practice facilitation in a cluster randomized stepped-wedge design trial to improve adherence to cardiovascular disease prevention guidelines: HealthyHearts NYC. Implement Sci. 2016 Jul 4;11(1):88. doi: 10.1186/s13012-016-0450-2. PMID 27377404